CLINICAL TRIAL: NCT06970574
Title: Comparative Study Between Intrathecal (Dexmedetomidine Versus Fentanyl) in Laparoscopic Cholecystectomies Under Spinal Anesthesia
Brief Title: Comparative Study Between Intrathecal (Dexmedetomidine Versus Fentanyl)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nehal Samir Esmail, Lecturer of Anesthesia, intensive care and pain management Faculty of Medicine, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: laparoscopic cholecystectomies
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2022-07

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Levobupivacaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 30 patients received 3.0 ml of heavy levo-bupivacaine with10 µg fentanyl (0.5 ml) to make 3.5 ml . All patients had been examined a day before surgery and will be kept fasting over-night, and received atropine 0.2 mg and ondansetron 8 mg intra venous as premedication. In the operation theater, patient's baseline pulse, blood pressure (BP), saturation, ETCO2, respiratory rate (RR), and electrocardiography (ECG) will be recordedand all will be preloaded with ringer lactate 15 ml/kg.
  Interventions: Drug: Levobupivacaine
- Group B (Active Comparator): About 30 patients received 3.0 ml of levo-bupivacaine along with dextmedetomidine 5 µg to make a total volume of 3.5 ml. All patients had been examined a day before surgery and will be kept fasting over-night, and received atropine 0.2 mg and ondansetron 8 mg intra venous as premedication. In the operation theater, patient's baseline pulse, blood pressure (BP), saturation, ETCO2, respiratory rate (RR), and electrocardiography (ECG) will be recordedand all will be preloaded with ringer lactate 15 ml/kg.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — to compare the clinical intraoperative effects of intrathecal administration of fentanyl in comparison with dexmedetomidine on shoulder tip pain in patients undergoing laparoscopic cholecystectomy.
  Other Names: fentanyl 50 mcg/ml; Dextmedetomidine

SUMMARY:
Laparoscopy is one of the procedures of choice for most of the elective abdominal surgeries performed preferably under endotracheal general anesthesia. With the technical advances that have been made, laparoscopic cholecystectomy is considered a procedure with a good safety profile that offers advantages over open cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopy is one of the procedures of choice for most of the elective abdominal surgeries performed preferably under endotracheal general anesthesia. With the technical advances that have been made, laparoscopic cholecystectomy is considered a procedure with a good safety profile that offers advantages over open cholecystectomy.

In past general anesthesia is considered the only choice of anesthesia for laparoscopy, but nowadays regional anesthesia in the form of spinal anesthesia, epidural anesthesia and or combined spinal epidural provide beneficial advantages over general anesthesia.

The most limiting factor for use of spinal anesthesia in laparoscopy is patient's discomfort with pneumo-peritoneum and the associated shoulder tip pain.

Spinal anesthesia is the most popular technique for lower abdominal surgeries as it is very economical and easy to administer. Various adjuvants have been added to intra-thecal local anesthetic agents. as Intrathecal α2 agonists when used as adjuncts potentiate the effect of local anesthetics and allows a decrease in required doses of local anesthetics.

Clonidine is a partial α2 agonist used intrathecally with well-established efficacy and safety. It prolongs the duration of motor and sensory spinal blockade when used along with local anesthetics. .

Dexmedetomidine is new highly selective α2 adrenoceptor agonist and has been approved by Food and Drug Administration as intravenous (IV) sedative and co-analgesic drug. Its α2/α1 selectivity is 8 times higher than clonidine.

many studies have been conducted the effect of intrathecal dexmedetomidine when combined with levobupivacaine in spinal anesthesia. However, not much literature is available regarding the use of intrathecal dexmedetomitine with levobupivacaine to reduce shoulder tip pain in laparoscopic cholecystectomies.

ELIGIBILITY:
Inclusion Criteria:

- 60 patients aged from 30 to 60 years of either sex with American Society of Anesthesiologists (ASA) grades I and II undergoing Elective laparoscopic cholecystectomies.

Exclusion Criteria:

* patients with ASA grade >II,
* Patients' refusal ,
* Patients using α2-adrenergic receptors antagonists, calcium channel blockers,
* angiotensin converting enzyme inhibitors ,
* Dysrhythmia ,
* Body weight more than 120 kg,
* spinal deformity ,
* History of allergy to the study drugs ,
* Pregnancy ,
* Coagulopathy ,
* Neurological disorders
* known contraindications to spinal anesthesia.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Effect of pneumoperitonum to shoulder pain | from 0 hours to 6 hours after the procedure
  Assessment of Intraoperative complaints of shoulder tip pain after carbon dioxide insufflation, using four grades [0, no pain; 1, mild pain but no need for analgesic; 2, moderate pain and need for analgesic; 3, severe pain and no response to analgesics (need for conversion to general anesthesia)]. And the severity will be observed using the 10 visual analogue scale where 0 meant no pain and 10 meant worst pain experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed hamody Hassan, Assist. Prof., Principal Investigator — Anesthesiology, Intensive care, and Pain Management, Faculty of Medicine, Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided